CLINICAL TRIAL: NCT01498172
Title: BCG Modulation of the recMAGE-A3 + AS15 ASCI Response in the Treatment of Patients With Non Muscle Invasive Bladder Cancer
Brief Title: BCG Modulation of the recMAGE-A3 + AS15 ASCI Response in the Treatment of Non Muscle Invasive Bladder Cancer (NMIBC) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Patrice Jichlinski (Other)
Collaborators: Ludwig Center for Cancer Research of Lausanne (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Patrice Jichlinski, Chief of Urology Department, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-68/11
Record Dates: First submitted 2011-12-06; First posted 2011-12-23 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Bladder Cancer
Keywords: Non muscle invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NMIBC at intermediate risk of progression (Experimental)
  Interventions: Biological: MAGE-A3 ASCI; Biological: BCG
- NMIBC at high risk of progression (Experimental)
  Interventions: Biological: MAGE-A3 ASCI; Biological: BCG
- NMIBC at low risk of progression (Experimental)
  Interventions: Biological: MAGE-A3 ASCI

INTERVENTIONS:
Biological: MAGE-A3 ASCI — 5 doses every 3 weeks
Biological: BCG — 1 intravesical dose /week for 6 weeks
  Other Names: Oncotice
  Arms: NMIBC at high risk of progression; NMIBC at intermediate risk of progression

SUMMARY:
In this study, the investigators would like to assess how intravesical BCG schedules after immunization of non muscle invasive bladder patients with the recMAGE-A3 protein, together with adjuvant AS15 (recMAGE-A3 + AS15 ASCI), may enhance innate and vaccine-specific T cell responses both systemically and locally in the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with histological confirmation of NMIBC
* Full recovery from surgery (TUR) from 1 to 6 weeks
* Karnofsky performance status of 60% or more
* Laboratory parameters for vital functions should be in the normal range
* Women of childbearing potential must use adequate contraception and have negative pregnancy test before and during the whole period of study treatment administration
* Male patients should avoid behaviors leading to child conception up to 2 months after administration of study treatment

Exclusion Criteria:

* Muscle invasive bladder cancer
* Metastatic disease to the central nervous system, for which other therapeutic options, including radiotherapy, may be available
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders)
* Any confirmed or suspected immunosuppressive or immunodeficient condition or potential immune-mediated diseases(Patients with vitiligo are not excluded to participate in the trial)
* History of severe allergic reactions to vaccines or unknown allergens
* Patients require concomitant chronic treatment with systemic corticosteroids or any other immunosuppressive agents.

The use of prednisone, or equivalent, <0.125 mg/kg/day (absolute maximum 10 mg/day), or inhaled corticosteroids or topical steroids is permitted

* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study agent
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability for immunological and clinical follow-up assessment
* For female patients of childbearing potential: positive urine or serum pregnancy test or lactating
* Known positive HIV test, HBV, HCV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Recording adverse events by assessment of vital signs, physical examination, haematology and blood chemistry to measure safety and tolerability | 6 months

SECONDARY OUTCOMES:
Flow cytometric analysis of type and number of immune cell types in urine | 6 months
Measurement of titers of antibodies against recMAGE-A3 in serum | 6 months
Assessment of disease recurrence by control cystoscopy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Jichlinski, MD, Principal Investigator — University Hospital Lausanne (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland